CLINICAL TRIAL: NCT07047521
Title: A Randomized, Double-Blind, Phase 3 Trial to Investigate the Immunogenicity and Safety of a New Formulation of Tetravalent Dengue Vaccine (TDV) Versus the Current Formulation of TDV in Healthy Adults (Aged 18-60 Years) in a Non-Endemic Area for Dengue
Brief Title: A Study on a New Tetravalent Dengue Vaccine (TDV) Formulation in Healthy Adults
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEN-322
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Dengue Fever
Keywords: Vaccine
MeSH Terms: conditions — Dengue | interventions — Dengue Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tetravalent Dengue Vaccine (TDV) (New) (Experimental): Participants will receive TDV (new formulation) dose 1, subcutaneous injection, once on Day 1 (first dose) and Day 90 (second dose).
  Interventions: Biological: Tetravalent Dengue Vaccine (TDV)
- Tetravalent Dengue Vaccine (TDV) (current) (Experimental): Participants will receive TDV (current approved formulation) 0.5 mL dose, subcutaneous injection, once on Day 1 (first dose) and Day 90 (second dose).
  Interventions: Biological: Tetravalent Dengue Vaccine (TDV)

INTERVENTIONS:
Biological: Tetravalent Dengue Vaccine (TDV) — TDV subcutaneous injection
  Other Names: TAK-003

SUMMARY:
Dengue fever is caused by an infection with the dengue virus. Vaccination with Dengue Tetravalent Vaccine (TDV) can help prevent dengue fever. The TDV in current formulation has been approved by health authorities in many countries around the world. The main aim of the study is to confirm that the TDV new formulation induces the similar immune response as approved TDV.

Healthy adults who live in an area in which dengue fever does not occur will receive 2 TDV vaccinations 3-months apart with either the new or the current TDV. Blood samples will be taken before and after the vaccinations. These are necessary to check how well the vaccine works to activate the immune system. During the study, participants will visit their study clinic 5 times.

ELIGIBILITY:
Inclusion Criteria

* Participant eligibility is determined according to the following criteria:
* Participant is aged 18 to 60 years at the time of entry into the trial.
* Participant is male or female.
* Participant is in good health at the time of entry into the trial, as determined by medical history, physical examination, and the clinical judgment of the investigator.
* Participant is immunologically naive to dengue, based on negative results for the detection of anti-DENV antibodies as documented by serological testing at screening.
* Participant has signed and dated a written informed consent form (ICF) and any required privacy authorization prior to the initiation of any trial procedures, and after the nature of the trial has been explained according to local regulatory requirements.
* Participant can comply with trial procedures and is available for the duration of follow-up.

Exclusion Criteria

* Participant has contraindication(s), warning(s), and/or precaution(s) applicable to vaccination with TDV as specified in the IB and/or approved product label in the participating country.
* Participant has a known hypersensitivity or allergy to any of the Dengue Tetravalent Vaccine (Live, Attenuated) (TDV) components (including excipients).
* Participant has behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, could interfere with the participant's ability to take part in the trial.
* Participant has a history of progressive or severe neurologic disorder, seizure disorder, or neuro-inflammatory disease (eg, Guillain-Barré syndrome).
* Participant has an illness or history of any illness that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the participant due to involvement in this trial.
* Participant has a known or suspected altered immunocompetence, including:

  1. Chronic administration of oral and/or parenteral steroids at doses considered sufficiently immunosuppressive (example, greater than and equal to [>=] 2 milligrams per kilograms [mg/kg] body weight/day prednisone [or equivalent] for >=14 consecutive days or >=20 mg/day prednisone [or equivalent] administered for >=14 consecutive days) within 60 days prior to Day 1 (Month [M] 0) (note: use of corticosteroids by inhaled, intranasal, intra-articular, bursal, tendon injection, or topical routes is allowed).
  2. Receipt of immunoglobulins and/or any blood products within the 3 months prior to Day 1 (M0) or planned administration during the trial.
  3. Receipt of immunostimulants within 60 days prior to Day 1 (M0).
  4. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Day 1 (M0).
  5. Human immunodeficiency virus (HIV) infection or HIV-related disease.
  6. Hepatitis B virus infection.
  7. Hepatitis C virus infection.
  8. Genetic immunodeficiency. 7. Participant has known or suspected abnormalities of splenic or thymic function.

     8. Participant has a known bleeding diathesis or any condition/medication that may be associated with a prolonged bleeding time.
* Participant has a serious chronic or progressive disease deemed to be preclusive to trial entry, that is, not medically stable according to the judgment of the investigator.
* Participant has a known previous infection with any flavivirus, including dengue, yellow fever, Japanese encephalitis, or tick-borne encephalitis viruses.
* Participant has previous or planned (during the trial conduct) vaccination against any flavivirus, including dengue (investigational or licensed vaccine), yellow fever viruses, Japanese encephalitis, or tick-borne encephalitis.
* Participant has a clinically significant active infection (as assessed by the investigator) or body temperature >= 38.0 degrees Celsius (°C) (>=100.4 degrees Fahrenhit [°F]) within 3 days of intended TDV administration.
* Participant has used antipyretics and/or analgesic medications within 24 hours prior to vaccination. The reason for their use (prophylaxis vs treatment) must be documented. Trial entry must be delayed to allow for a full 24 hours to have passed since last use of antipyretics and/or analgesic medications.
* Participant has a history of substance or alcohol abuse within the past 2 years.
* Female participants who are pregnant (ie, a positive or indeterminate pregnancy test).
* Female participants who are breastfeeding.
* Female participants of childbearing potential1 who are sexually active and who have not used any of the acceptable contraceptive methods2 for at least 2 months prior to Day 1 (M0).
* Female participants of childbearing potential1 who are sexually active with a non-sterilized male partner and refuse to use an acceptable contraceptive method up to 6 weeks post second TDV vaccination on Day 90 (M3), or who are planning to donate ova up to 6 weeks each post first (on Day 1 [M0]) and post second (on Day 90 [M3]) TDV administration.
* Non-sterilized male participants who are sexually active with a female partner of childbearing potential1 and refuse to use a barrier method 4 of contraception up to 6 weeks each post first (on Day 1 [M0]) and post second (on Day 90 [M3]) TDV administration, or who are planning to donate sperm during these periods.
* Participant has received any of the following:

  1. A licensed vaccine within 14 days (for inactivated or mRNA vaccines) or 28 days (for live or vector-based [if vector amplifies in body] vaccines) prior to TDV administration.
  2. A vaccine authorized for emergency use within 28 days prior to TDV administration.
* Participant is scheduled to receive any vaccine within 28 days after TDV administration.
* Participant is participating in any clinical trial with another investigational product 30 days prior to Day 1 (M0) or intending to participate in another clinical trial at any time during the conduct of this trial.
* Participant has taken part in any clinical trial of a dengue or other flavivirus (example, West Nile virus, Japanese encephalitis) candidate vaccine, except if it is known that the participant received placebo in those trials.
* Participant is planning to donate blood, organs, or tissues up to 6 weeks post second vaccination on Day 90 (M3).
* Participant or their first-degree relatives are involved in the trial conduct.
* Participant identified as an employee of the investigator or trial center, with direct involvement in the proposed trial or other trials under the direction of that investigator or trial center.
* Participant has lived in a dengue-endemic area for >=3 months.
* Participant has planned travel (during trial conduct) to any endemic area for dengue and other flaviviruses.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 496 (Actual)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titers (GMTs) of Neutralizing Antibodies (By MNT) Against Each of the 4 Dengue Serotypes at Day 120 In the TDV (New) And TDV (Current) Groups | At Day 120
  GMTs of neutralizing antibodies will be measured by microneutralization test 50% [MNT50] for each of the 4 Dengue Serotypes. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. GMTs of neutralizing antibodies (by MNT) against each of the 4 dengue serotypes at Day 120 in the TDV (new) and TDV (current) groups will be reported.

SECONDARY OUTCOMES:
GMTs of Neutralizing Antibodies (By MNT) Against Each of the 4 Dengue Serotypes at Day 270 In the TDV (New) And TDV (Current) Groups | At Day 270
  GMTs of neutralizing antibodies will be measured by microneutralization test 50% [MNT50] for each of the 4 Dengue Serotypes. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. GMTs of neutralizing antibodies (by MNT) against each of the 4 dengue serotypes at Day 270 in the TDV (new) and TDV (current) groups will be reported.
Seropositivity Rates Against Each of the 4 Dengue Serotypes at Day 120 And Day 270 In the TDV (New) And TDV (Current) Groups | At Days 120 and 270
  Seropositivity rate is defined the percentage of participants seropositive, was derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a neutralizing titer >=10 against each of the four dengue virus serotypes. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Seropositivity Rates Against Multiple (2, 3 or 4) Dengue Virus Serotypes at Day 120 And Day 270 In the TDV (New) And TDV (Current) Groups | At Days 120 and 270
  Seropositivity rate is defined the percentage of participants seropositive, was derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a neutralizing titer >=10 against multiple (2, 3, or 4) dengue virus serotypes. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 days Post Vaccination (Overall and by Severity) | Within 7 Days post-vaccination at Day 1 and Day 90
  Solicited local AEs are injection site pain/tenderness, erythema, and swelling at the vaccination site. All solicited AEs at the injection site will be considered related to the study vaccine administration. The AEs of severity will be graded by investigator as Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants With Solicited Systemic AEs for 14 days Post Vaccination (Overall and by Severity) | Within 14 days post-vaccination at Day 1 and Day 90
  Solicited systemic AEs include fever (body temperature greater than or equal to [>=] 38-degree Celsius [C], drowsiness, irritability/fussiness and loss of appetite. The AEs of severity will be graded by investigator as Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants With Any Unsolicited Adverse Events (AEs) for 28 days Post Vaccination | Within 28 days post-vaccination at Day 1 and Day 90
  An unsolicited AE is any AE reported by the participant that is not specified as a solicited AE or is specified as a solicited AE but starts outside the period for reporting a solicited AE (that is, 7 days and 14 days in total including the day IMP administration).
Percentage of Participants With Serious Adverse Events (SAEs) Throughout the Study | From first vaccination (Day 1) through end of study (Day 270)
  An SAE was defined as any untoward medical occurrence or effect that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically important due to other reasons than the above mentioned criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- Australia (5):
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - Emeritus Research Sydney, Botany, New South Wales
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - Veritus Research, Bayswater, Victoria
  - Emeritus Research Camberwell (Melbourne), Camberwell, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/70cdfca5c83743cf??page=1&idFilter=DEN-322